CLINICAL TRIAL: NCT00080288
Title: A 12 Week, Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of CEP 10953 (150 mg) as Treatment for Adults With Excessive Sleepiness Associated With Chronic Shift Work Sleep Disorder
Brief Title: Safety/Efficacy Study With Armodafinil (CEP-10953) in Treatment of Excessive Sleepiness Associated With Chronic SWSD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C10953/3022/CM/MN
Record Dates: First submitted 2004-03-25; First posted 2004-03-29 (Estimated); Results first posted 2009-09-23 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Excessive Sleepiness; Shift Work Sleep Disorder
Keywords: Excessive Sleepiness; Chronic Shift Work Sleep Disorder; Chronic SWSD; Circadian Rhythm Disorder; Shift Worker; Cephalon; Cephalon, Inc; Nuvigil
MeSH Terms: conditions — Disorders of Excessive Somnolence; Sleep Disorders, Circadian Rhythm; Chronobiology Disorders | interventions — Modafinil

ARMS (2):
- 1 (Experimental): Armodafinil 150 mg/day
  Interventions: Drug: Armodafinil 150 mg/day
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Armodafinil 150 mg/day — Armodafinil 150 mg taken 30 minutes to 1 hour before the start of the night shift, but no later than 2300, only on nights worked.
  Arms: 1
Drug: Placebo — Matching placebo tablets once daily
  Arms: 2

SUMMARY:
The primary objective of this study is to determine whether treatment with Armodafinil (CEP-10953) is more effective than placebo treatment for patients with excessive sleepiness associated with chronic shift work sleep disorder (SWSD) by measuring mean sleep latency from the Multiple Sleep Latency Test (MSLT) (20 minutes) (average of 4 naps at 0200, 0400, 0600, and 0800) and by Clinical Global Impression of Change (CGI-C) ratings.

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if all of the following criteria are met:

* Written informed consent is obtained.
* The patient is an outpatient, man or woman of any ethnic origin, 18 to 65 years of age (inclusive).
* The patient has a complaint of excessive sleepiness.
* The patient has a diagnosis of SWSD according to International Classification of Sleep Disorders (ICSD) criteria, and must have had excessive sleepiness during night shifts for at least 3 months.
* The patient must work at least 5 night shifts per month, of which at least 3 nights are consecutive, and plan to maintain this schedule.
* The patient must work night shifts that include at least 6 hours between 2200 and 0800 and be no longer than 12 hours in duration.
* The patient is in good health as determined by a medical and psychiatric history, physical examination, ECG, and serum chemistry and hematology.
* Women must be surgically sterile, 2 years postmenopausal, or, if of child-bearing potential, using a medically accepted method of birth control (ie, barrier method with spermicide, steroidal contraceptive, or intrauterine device [IUD]) and agree to continued use of this method for the duration of the study. Steroidal contraceptives must be used with a barrier method while taking the study drug and for at least a full cycle after discontinuation of the study drug.
* The patient has a mean sleep latency of 6 minutes or less as determined by the MSLT
* The patient has a CGI-S rating as it pertains to sleepiness during night shifts including the commute to and from work.
* The patient does not have any medical or psychiatric disorders that could account for the excessive sleepiness during the night shift.
* The patient is able to complete self rating scales and computer-based testing.
* The patient is willing and able to comply with study restrictions and to attend regularly scheduled clinic visits as specified in this protocol.

Exclusion Criteria:

Patients are excluded from participating in this study if 1 or more of the following criteria are met:

* has any clinically significant, uncontrolled medical or psychiatric conditions (treated or untreated)
* has a probable diagnosis of a current sleep disorder other than SWSD
* consumes caffeine including coffee, tea and/or other caffeine containing beverages or food averaging more than 600 mg of caffeine per day
* used any prescription drugs disallowed by the protocol or clinically significant use of over the-counter (OTC) drugs within 7 days before the screening/baseline visit
* has a history of alcohol, narcotic, or any other drug abuse as defined by the Diagnostic and Statistical Manual of Mental Disorders of the American Psychiatric Association, 4th Edition (DSM IV)
* has a positive urine drug screen (UDS) at the screening visit
* has a clinically significant deviation from normal in the physical examination
* is a pregnant or lactating woman. (Any woman becoming pregnant during the study will be withdrawn from the study.)
* has used an investigational drug within 1 month before the screening visit
* has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery)
* has a known clinically significant drug sensitivity to stimulants or modafinil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2004-03; Study Completion 2004-12

REFERENCES:
- [Derived] Czeisler CA, Walsh JK, Wesnes KA, Arora S, Roth T. Armodafinil for treatment of excessive sleepiness associated with shift work disorder: a randomized controlled study. Mayo Clin Proc. 2009 Nov;84(11):958-72. doi: 10.1016/S0025-6196(11)60666-6. PMID 19880686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 centers (37 in US, 5 in Canada). First patient enrolled: 2 April 2004/ Last patient last visit: 23 December 2004
Pre-assignment Details: 9 participants (3 female ; 6 male) withdrew after randomization but prior to receiving study drug. These 9 patients are included in the Participant Flow table below.
Period: Overall Study
Arm/Group | Armodafinil 150 mg/Day | Placebo
Started | 127 | 127
Completed | 97 | 89
Not Completed | 30 | 38
Not completed — Adverse Event | 7 | 4
Not completed — Lost to Follow-up | 3 | 5
Not completed — Physician Decision | 6 | 2
Not completed — Withdrawal by Subject | 3 | 16
Not completed — Miscellaneous | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil 150 mg/Day | Placebo | Total
Number analyzed (Participants) | 127 | 127 | 254
Age Categorical [Number; unit: participants] — 9 participants (3 female ; 6 male) withdrew after randomization but prior to receiving study drug
  participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 123 | 122 | 245
    >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.9 (10.75) | 40.3 (10.76) | 39.6 (10.76)
Gender [Number; unit: participants] — 9 participants (3 female ; 6 male) withdrew after randomization but prior to receiving study drug
  participants
    Female | 57 | 58 | 115
    Male | 66 | 64 | 130
Region of Enrollment [Number; unit: participants]
  United States | 117 | 117 | 234
  Canada | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Multiple Sleep Latency Test (MSLT)
Description: The Multiple Sleep Latency Test (MSLT) is an objective assessment of sleepiness that measures the ability of a subject to remain awake. Long latencies to sleep are indicative of a patient's ability to remain awake. Mean sleep latency from MSLT was measured for five 20-minute (maximum) MSLT naps performed at scheduled visits (2400 [midnight], 0200, 0400, 0600, and 0800).The MSLT was administered at weeks 4, 8, and 12. The primary efficacy variable was the mean change from the baseline assessment in MSLT sleep latency as assessed at week 12 (or last postbaseline visit).
Time Frame: up to 12 weeks
Population: Safety Analysis set of 245 total patients: 9 participants withdrew after randomization but prior to receiving study drug
  Full Analysis set of 216 total patients: 29 patients that had withdrawn from the study were non-evaluable for efficacy.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 112 | 104
Minutes | 3.1 (4.46) | 0.4 (2.87)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Assumption: both primary treatment comparisons would be with a 2 sided test at an alpha level of 0.05; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 2.7, 95% CI [1.67 to 3.69]

2. Primary Outcome: Clinical Global Impression of Change (CGI-C)
Description: Number of participants who had at least minimal improvement in CGI-C ratings at Week 12 or last post-baseline visit. The CGI-C uses the following categories and scoring assignments: 1=Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; and 7=Very much worse. Severity of illness was assessed at baseline by the CGI-S, which consists of the following categories: 1=Normal (shows no signs of illness); 2=Borderline ill; 3=Mildly (Slightly) ill; 4=Moderately ill; 5=Markedly ill; 6=Severely ill; and 7=Among the most extremely ill patients.
Time Frame: up to 12 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 112 | 104
Participants | 112 | 104
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Assumption: both primary treatment comparisons would be with a 2 sided test at an alpha level of 0.05; Test type: Superiority or Other; p = 0.0010, Cochran-Mantel-Haenszel; The p value for each treatment group is for the comparison of that treatment group to the placebo treatment group. Adjusted for country

ADVERSE EVENTS:
Arm/Group | Armodafinil 150 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 1/123 | 1/122
Other Adverse Events (participants affected / at risk) | 28/123 | 18/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 150 mg/Day (N=123) | Placebo (N=122)
Meningitis viral (Infections and infestations) | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 150 mg/Day (N=123) | Placebo (N=122)
Nausea (Gastrointestinal disorders) | 9 | 4
Nasopharyngitis (Infections and infestations) | 7 | 4
Headache (Nervous system disorders) | 15 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days